CLINICAL TRIAL: NCT03983369
Title: Multicenter Double Blind Randomized Placebo-controlled Trial Assessing the Efficacy of Low-level Laser Therapy in the Prevention of Chemotherapy-induced Mucositis in Children and Young Adults
Brief Title: Low-level Laser Therapy in the Prevention of Chemotherapy-induced Mucositis in Children and Young Adults
Acronym: MUCILA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-A03041-52; 2017/2640 (Other: CSET number)
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mucositis Oral
MeSH Terms: conditions — Stomatitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This is a superiority trial, multicenter, prospective, randomized in two parallel groups (containing a placebo control group) and a double-blind assessment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Multicenter randomized double blind placebo-controlled trial stratified according to the type of chemotherapy (Stratum A and B) and by center. Patients will be randomized in two parallel groups: preventive treatment with LLLT ("Laser" group) or a control group with a placebo intervention ("Placebo" group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preventive treatment with LLLT ("Laser" group) (Experimental)
  Interventions: Device: Low-Level Laser Therapy
- control group with a placebo intervention (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Low-Level Laser Therapy — The LLL used is the K-Laser Cube 3. The LLL is an athermal laser beam of low power, equipped with a placebo function (dummy imitating beam laser light, emitted by the same device but without physiological effect).
  Arms: preventive treatment with LLLT ("Laser" group)
Other: Placebo — Placebo
  Arms: control group with a placebo intervention

SUMMARY:
To assess the efficacy of preventive Low-Level Laser Therapy (LLLT) for reducing the incidence of WHO's grade 3-4 oral mucositis in children and young adults receiving chemotherapy regimens associated with a high rate of mucositis: conventional chemotherapy or High Dose Chemotherapy (HDC) conditioning regimens with Hematological Stem Cell Transplantation (HSCT).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 4 and ≤ 25 years
2. No mucositis or other mouth lesions at the beginning of chemotherapy that could prevent the laser session and chemotherapy
3. Cooperative patient, able to wear black glasses and to sit with his open mouth during laser session
4. Patients treated in one of the SFCE centers that participate to the study
5. Patients undergoing chemotherapy course with high risk of severe mucositis :

   1. high-dose chemotherapy with hematological stem cell transplantation (stratum A) including but not limited to 8 HDC conditioning regimens for solid tumors intensive treatment (Busilvex-Melphalan, VP16-Thiotepa, BAM, BEAM, Thiotepa 900mg/m^2, Carboplatine-Thiotepa (typical teratoid rhabdoid tumor or medulloblastoma), VP16-Carboplatine-Thiotepa, Endoxan-Busilvex and VP16 - Melphalan) and 5 myeloablative conditioning regimens (for example : TBI-VP16, Busilvex-Endoxan-Thiotepa, Busilvex-Endoxan+/-Melphalan and Thiotepa-Busulfan-Fludarabine),
   2. Conventional chemotherapy courses (stratum B) but not limited to COPADM (B lymphoma), CAV/ICE (plexus choroid carcinoma or B lymphoma), Head start induction course (medulloblastoma), N6 course (neuroblastoma), VIDE or VCD (Ewing sarcoma), API/AP (osteosarcoma), Cyclophosphamide and Doxorubicine (nephroblastoma), PLADO/Carboplatine and Doxorubicine (hepatoblastoma), IVADo (rhabdomyosarcoma), induction and consolidation of the Myechild protocol (Cytarabine/Mithoxantrone Fludarabine Aractine +/- Darubicine) (acute myeloid leukemia) and 5FU-cisplatine (undifferentiated carcinoma of nasopharyngeal),
   3. Others courses of chemotherapy (stratum A or B) which may cause mucositis can be considered (please refer to the non-inclusion criterion n° 5 to see the prohibited chemotherapy list). In this case, the coordinating investigator approval is required.
6. Women of childbearing potential must have a negative serum β-HCG pregnancy test prior to the administration of the first laser treatment.
7. French speaking patients
8. Patient and/or parents/legal representatives should understand, sign, and date the written informed consent form prior to any protocol specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
9. Patients must be affiliated to a social security regimen or beneficiary of the same

NB : all patients who respect all the eligibility criteria are recruitable even if the patient haven't a cancer (Patients undergoing a chemotherapy with high risk of severe mucositis for another clinical reason than cancer).

Exclusion Criteria:

1. Treatment by opioids on daily basis
2. Orthodontic appliance
3. Pregnant or breastfeeding young ladies or women
4. Patients with cognitive disorder who could not self-evaluate his pain or with a mucositis difficult to evaluate
5. None of this chemotherapy is allowed : Methotrexate, VA or VAD (nephroblastoma), Carboplatine - Etoposide (3 or 5 days), Temozolomide single agent or in combination with Topotecan/Irinotecan or Bevacizumab, Gemzar, Taxotere, Ifosfamide - Etoposide (Ewing sarcoma), OEPA, COPDAC, IgEV (Hodgkin lymphoma)

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 315 (Estimated)
Dates: Start 2018-08-29 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of grade 3-4 mucositis | assessed at day 12 ± 2 days after initiation of chemotherapy

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Gustave Roussy, Villejuif, Val de Marne
  - Centre Oscar Lambret, Lille
  - Hôpital Robert Debré, Paris
  - Institut Curie, Paris
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided